CLINICAL TRIAL: NCT00681655
Title: GABRA2 and the Pharmacokinetics of Risk for Alcoholism (GPRA)
Acronym: GPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sean O'Connor, Professor, Department of Psychiatry and Biomedical Engineering, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: O'CONNOR_AA007611-18; P60AA007611 (NIH)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Two session, within subjects, single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Responses to alcohol (Experimental): Each subject completed a total of 2 2.8 hr-long clamping sessions.Within each session, procedures differed only by the content of the infusate. In one session, 6% ethanol was infused. In the other session, only vehicle was infused, quantifying the placebo response for every subject. The order of alcohol or placebo sessions was counterbalanced; subjects were blind to which session was which; sessions were scheduled to occur about 2 weeks apart. Measures were collected before, and at beginning and end of infusion, and included subjective perceptions, EMG, EEG, stop-signal performance, eye movements, and auditory responses. Design allowed analysis of effect of alcohol vs placebo, initial effect of alcohol and acute tolerance to alcohol.
  Interventions: Other: Alcohol; Other: Placebo

INTERVENTIONS:
Other: Alcohol — Alcohol (6% in saline vehicle) infused for 2.8 hour long clamping session (Breath alcohol level maintained at 60 mg/dL throughout).
Other: Placebo — Placebo (saline vehicle) infused for 2.8 hour long session.

SUMMARY:
This study will assess whether the presence of a particular form of a gene, GABRA2, affects the functional responses of the human brain to alcohol administration and will evaluate that relationship in the context of factors known to increase the risk for future alcoholism.

DETAILED DESCRIPTION:
Each subject completed a total of 2 2.8 hr-long clamping sessions.Within each session, procedures differed only by the content of the infusate. In one session, 6% ethanol was infused. In the other session, only vehicle was infused, quantifying the placebo response for every subject. The order of alcohol or placebo sessions was counterbalanced; subjects were blind to which session was which; sessions were scheduled to occur approximately 2 weeks apart. Measures were collected before, and at beginning and end of infusion, and included subjective perceptions, EMG, EEG, stop-signal performance, eye movements, and auditory responses. Design allowed analysis of effect of alcohol vs placebo, initial effect of alcohol and acute tolerance to alcohol.

ELIGIBILITY:
Inclusion Criteria:

* European American male and females between 21-27 years of age.
* Good health as determined by medical history, physical exam, and laboratory tests.
* Females must have a negative urine pregnancy (hCG) test at the start of each study session.
* People who consume 0.10 standard drinks per week (12 g-ethanol) per liter of total body water when averaged over the preceding month, or more, OR who have consumed more than 0.10 standard drinks per liter of total body water on any one occasion in the last month.

Exclusion Criteria:

* Inability to read or comprehend eighth grade English.
* Inability to hear or comprehend verbal instructions, or inability or unwillingness to cooperate with the procedures required for the study.
* Inability to resolve 2 dots, each 2 mm in diameter with centers placed 5 mm apart on a card placed 20 inches from the bridge of the nose, or the need to wear eyeglasses to do so.
* Current or prior history of any serious disease, including head trauma causing loss of consciousness, cancer, CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or alcohol or drug dependence, but not alcohol abuse or nicotine dependence.
* Positive hepatitis or HIV test at screening, provided subject consented to these tests.
* Current or prior history of alcohol-induced flushing reactions.
* Current diagnosis of Axis-I psychiatric illness.
* Positive result on urine drug screen obtained at the face-to-face interview.
* Pregnancy, as determined by urine HcG on each day of laboratory testing, or intention to become pregnant for women.
* Use of medications known to interact with alcohol within 2 weeks of the study.

Ages: 21 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2008-05; Primary Completion 2012-04-14 (Actual); Study Completion 2012-04-14 (Actual)

PRIMARY OUTCOMES:
Effect of GABRA2 SNP status on AUD risk | Both session responses and lifetime traits will be included in analysis
  Results will assess the effect of GABRA2 SNPs on responses to alcohol and traits related to alcoholism risk

SECONDARY OUTCOMES:
Acute tolerance to alcohol | Within 3 hour session
  Comparison of measures taken during the initial hour of the clamp with the same measures taken during the 3rd hour of the alcohol clamp.
Initial response to alcohol | Within 3 hour session
  Comparison of measures taken during baseline with the same measures taken during the initial hour of the alcohol clamp.
Responses to alcohol vs placebo | Within 3 hour session
  Measures taken during the alcohol session will either be compared to those taken during placebo, or in some cases measures taken during the alcohol session will be corrected for placebo effects by subtracting placebo responses from alcohol responses

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Plawecki, M.D., Study Director — Indiana University School of Medicine; Sean J. O'Connor, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing will be considered on a case by case basis. No sharing of HIPPA sensitive data will be allowed.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: While lab analyses are ongoing, data is available on request
Access Criteria: Data access requests will be reviewed by the investigators. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Result] Kosobud AE, Wetherill L, Plawecki MH, Kareken DA, Liang T, Nurnberger JL, Windisch K, Xuei X, Edenberg HJ, Foroud TM, O'Connor SJ. Adaptation of Subjective Responses to Alcohol is Affected by an Interaction of GABRA2 Genotype and Recent Drinking. Alcohol Clin Exp Res. 2015 Jul;39(7):1148-57. doi: 10.1111/acer.12749. Epub 2015 Jun 19. PMID 26087834
- [Result] Plawecki MH, Windisch KA, Wetherill L, Kosobud AEK, Dzemidzic M, Kareken DA, O'Connor SJ. Alcohol affects the P3 component of an adaptive stop signal task ERP. Alcohol. 2018 Aug;70:1-10. doi: 10.1016/j.alcohol.2017.08.012. Epub 2017 Aug 31. PMID 29705707